CLINICAL TRIAL: NCT06627751
Title: Phase II Clinical Trial of Mezigdomide/Carfilzomib/Dexamethasone (MeziKD) in Patients With Relapsed or Refractory Multiple Myeloma (MM) With Extramedullary Disease (EMD)
Brief Title: Mezigdomide, Carfilzomib, and Dexamethasone for the Treatment of Relapsed or Refractory Multiple Myeloma in Patients With Extramedullary Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-3576824
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Extramedullary Disease in Multiple Myeloma; Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate; dexamethasone acetate; dexamethasone 21-phosphate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment - MeziKD (Experimental): Patients receive mezigdomide PO QD on days 1-21 of each cycle, carfilzomib IV over 30 minutes on days 1, 8, and 15 of each cycle, and dexamethasone PO on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. After 6 cycles of study treatment, patients showing a response to therapy may continue the treatment regimen as part of standard of care per physician's discretion. Additionally, patients undergo ECHO, PET/CT, MRI, CT guided tumor biopsy, bone marrow aspiration and biopsy, and blood and saliva sample collection throughout the study,
  Interventions: Biological: Mezigdomide; Drug: Carfilzomib; Drug: Dexamethasone; Procedure: Echocardiography; Procedure: Positron Emission Tomography; Procedure: Computed Tomography; Procedure: Computed Tomography Assisted Biopsy; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Biospecimen Collection

INTERVENTIONS:
Biological: Mezigdomide — Given PO
  Other Names: BMS 986348; CC-92480
Drug: Carfilzomib — Given IV
  Other Names: CFZ
Drug: Dexamethasone — Given PO
  Other Names: Adexone; Baycadron; Cortidexason; Decadron; Dekacort; Fortecortin; Gammacorten; Hexadecadrol; Loverine; Millicorten; Orgadrone; Spersadex; TaperDex; Visumetazone
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: PET; PET scan
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan
Procedure: Computed Tomography Assisted Biopsy — Undergo CT guided tumor Biopsy
  Other Names: CT Assisted Biopsy
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
Procedure: Biospecimen Collection — Undergo blood and saliva sample collection
  Other Names: Biological Sample Collection

SUMMARY:
This phase II trial studies how well mezigdomide/carfilzomib/dexamethasone (MeziKD) works in treating patients with multiple myeloma (MM) that has come back after a period of improvement (relapsed) or that does not respond to treatment (refractory) and have tumors from myeloma cells outside the bone marrow in the soft tissues or organs of the body (extramedullary disease [EMD]). Mezigdomide blocks important processes in myeloma cells and may lead to modulation of the immune system, including activation of T-lymphocytes, and downregulation of the activity of other proteins, some of which play key roles in the proliferation of certain cancer cell types. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Dexamethasone is a type of corticosteroid and is used to kill myeloma cells. It is used with other drugs to treat multiple myeloma. Giving MeziKD may kill more cancer cells in patients with relapsed/refractory multiple myeloma (RRMM) with EMD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* RRMM patients with one or more prior lines of therapy with at least one ES or PS lesion that is accessible to a biopsy. Accessibility will be assessed by the MM tumor board
* Measurable disease meeting at least one of the following:

  * Serum M-protein ≥1 g/dL
  * Urine M-protein ≥200 mg/24 h
  * Serum FLC assay: involved FLC level ≥10 mg/dL provided serum FLC ratio is abnormal
  * Up to 10 patients without measurable disease can be enrolled but screening imaging and/or bone marrow biopsy have to confirm RRMM. Follow-up response assessment will be performed with imaging using RECIST 1.1 and Deauville Criteria and bone marrow biopsies
* Absolute neutrophil count: ≥ 1 x 10^9/L
* Platelets: ≥ 75 x 10^9/L
* Total bilirubin: ≤ 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]): ≤ 3 x ULN
* Renal function: Estimated creatinine clearance ≥ 30 mL/min (Cockroft-Gault)
* Adequate cardiac pump function with a left ventricular ejection fraction of ≥ 40%
* Women of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for at least 28 days after the last dose of mezigdomide or 6 months after the last dose of carfilzomib. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Male patients (non-vasectomized) must agree to use contraception during the treatment period and for at least 28 days after the last dose of mezigdomide or 3 months after the last dose of carfilzomib and refrain from donating sperm during this period
* Participant must understand the investigational nature of this study and sign an independent ethics committee/institutional review board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Participant has a history of anaphylaxis or hypersensitivity to thalidomide, lenalidomide, pomalidomide (including ≥ grade 3 rash during prior thalidomide, lenalidomide, or pomalidomide therapy), carfilzomib or dexamethasone, any cereblon E3 ligase modulators (CELMoD) agents, or the excipients contained in the formulations, or participant has any contraindications per local prescribing information
* Administration of strong CYP3A modulators or proton-pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, pantoprazole, rabeprazole) within 2 weeks of starting study intervention
* Participant is unable or unwilling to undergo protocol required thromboembolism prophylaxis
* Patient has evidence of mucosal or internal bleeding and/or is platelet transfusion refractory
* Any medical conditions that, in the investigator's opinion, would impose excessive risk to the patient or would adversely affect his/her participation in this study
* Known active infection requiring parenteral or oral anti-infective treatment within the past 14 days
* Participant has a history of prior malignancy other than MM, except if the participant has been free of disease for ≥ 3 years or the participant had 1 of the following noninvasive malignancies treated with curative intent without known recurrence:

  * Basal or squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix or breast
  * Stage 1 bladder cancer
  * Incidental histological findings of localized prostate cancer such as tumor stage 1a or 1b (T1a or T1b) using the tumor, nodes, and metastasis (TNM) classification of malignant tumors OR prostate cancer that has been treated with curative intent
* Other ongoing anti-myeloma therapy. Patients may be receiving concomitant therapy with bisphosphonates and low dose corticosteroids for symptom management and comorbid conditions. Doses of corticosteroid should be stable for at least 7 days prior to patient registration
* Pregnant or breast-feeding females
* Serious psychiatric illness, active alcoholism, or drug addiction that may hinder or confuse follow-up evaluation
* Known active HIV or hepatitis B or C viral infection
* Known history of HIV infection
* Systemic amyloidosis or POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein [M-protein] and skin changes)
* Prior peripheral stem cell transplant within 12 weeks of study enrollment
* Radiotherapy within 14 days prior to cycle 1 day 1. However, if the radiation portal covered ≤ 5% of the bone marrow reserve, the patient may be enrolled irrespective of the end date of radiotherapy
* Known intolerance to steroid therapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, severe cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Carfilzomib-refractory in the most recent line of therapy
* Prior treatment with mezigdomide
* Contraindication against conscious sedation
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | At the end of cycle 6 (each cycle is 28 days).
  Will be assessed in patients with serologically measurable disease. Will be defined as the percentage of patients with an objective response of partial response (PWR) or better by International Myeloma Working Group criteria on 2 consecutive evaluations among the eligible patients who began protocol treatment. Will be evaluated using a one-sided Binomial test and a 90% credible region for the overall response rate will be constructed using Jeffrey's prior method
Clinical benefit rate | At the end of cycle 6 (each cycle is 28 days)
  Will be assessed in patients with non- or oligo-secretory disease. Clinical benefit rate is the percentage of patients who remain progression-free and on protocol treatment for at least 6 months among the eligible patients who began protocol treatment. A 90% binomial credible region will be constructed for the clinical benefit rate using Jeffrey's prior method.

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 30 days after last dose of study drug
  As per Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0: type, frequency, seriousness, severity and relationship of AEs to mezigdomide and carfilzomib/dexamethasone. For each patient cohort, the AEs reported will be graded and an attribution assigned using CTCAE v5.0. For each patient, the maximum grade of each AE will be determined and the frequency of each AE by max grade will be tabulated for each cohort.
Duration of response | From the first documentation of response (≥ PR) to the first documentation of progressive disease or death, assessed up to 3 years
  For those with and without serologically measurable disease, the DOR will be estimated by Kaplan-Meier method. Estimates of the median will be obtained with 90% confidence intervals
Progression Free survival | Time from first dose of mezigdomide to disease progression or death from any cause, whichever occurs first, assessed up to 3 years
  At screening, after 3 cycles of treatment (or progression, whichever occurs first), after 6 cycles of treatment, and then every 6 months for 3 years or until progression, start of a new therapy, or death (whichever occurs first)
Overall Survival | Time from first dose of mezigdomide to death from any cause, assessed up to 3 years
  At screening, after 3 cycles of treatment (or progression, whichever occurs first), after 6 cycles of treatment, and then every 6 months for 3 years or until progression, start of a new therapy, or death (whichever occurs first)
Imaging Response | At screening, after 3 cycles of treatment (or progression, whichever occurs first), after 6 cycles of treatment, and then every 6 months for 3 years or until progression, start of a new therapy, or death (whichever occurs first)
  Will be assessed in those without serologically measurable disease using positron emission tomography/computed tomography and magnetic resonance imaging. Will be assessed using Response Evaluation Criteria in Solid Tumors v1.1 and Deauville criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hillengass, MD, Principal Investigator — Roswell Park Comprehensive Cancer Center
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States